CLINICAL TRIAL: NCT04106596
Title: Immunogenetic Characteristics in Autoimmune Encephalitis and Related Disorders: HLA Analysis
Brief Title: HLA Analysis in Autoimmune Encephalitis and Related Disorders
Acronym: ICARE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ICARE
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Autoimmune Encephalitis; Imbic Encephalitis; Autoimmune Cerebellar Ataxia; Stiff-person Syndrome
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Stiff-Person Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood collected at diagnosis time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with antibodies against LGI1: This is a non-interventional study involving biological samples (DNA). Samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL)/NeuroBioTec (including tissue, cells or biological fluids) and genetic analysis for research purposes (e.g. involving genes related to the disease for which the patient was followed). Additionally, patients will be informed about the present study.
- Patients with antibodies against CASPR2: This is a non-interventional study involving biological samples (DNA). Samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL)/NeuroBioTec (including tissue, cells or biological fluids) and genetic analysis for research purposes (e.g. involving genes related to the disease for which the patient was followed). Additionally, patients will be informed about the present study.
- Patients with antibodies against GAD: This is a non-interventional study involving biological samples (DNA). Samples are already stored in biobank repositories and collected as part of "good clinical practice" in the diagnostic process of patients with suspected autoimmune encephalitis, meaning that the standard diagnostic and therapeutic approaches will not be altered in the selected study population. Patients have already gave explicit written consent for biological specimens sampling and storage at the "Centre de Ressources Biologiques des Hospices Civils de Lyon" (CRB-HCL)/NeuroBioTec (including tissue, cells or biological fluids) and genetic analysis for research purposes (e.g. involving genes related to the disease for which the patient was followed). Additionally, patients will be informed about the present study.

SUMMARY:
Autoimmune encephalitis (AE) are characterized by subacute onset of memory deficits, altered mental status or psychiatric symptoms, frequently associated with seizures, inflammatory cerebrospinal fluid and in cases with prominent limbic involvement, typical magnetic resonance imaging. Several autoantibodies (Ab) may be detected in AE, although its detection is not mandatory to establish a diagnosis. These Ab mainly recognize different synaptic and cell-surface proteins in the central nervous system, and are thought to be pathogenic as they alter the normal location or function of its antigens.

The primary trigger of the immune response is unknown for most of AE. In addition to acquired susceptibility, genetic predisposition may also be important in the pathogenesis of AE. Human leukocyte antigen (HLA) is the genetic factor most frequently associated with autoimmune diseases, due to its genetic complexity and key role in the adaptive immune response. The aim of the study is to describe HLA profile in three groups of autoimmune encephalitis and related disorders: anti-LGI1, anti-CASPR2 and anti-GAD neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of anti-LGI1, anti-CASPR2 or anti-GAD antibodies in serum or cerebrospinal fluid;
2. Clinical picture compatible with the detected antibody (limbic encephalitis in anti-LGI1; limbic encephalitis, neuromyotonia or Morvan's syndrome in anti-CASPR2; limbic encephalitis, cerebellar ataxia or stiff-person syndrome in anti-GAD

Exclusion Criteria:

- Absence of complete clinicobiological data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with autoimmune encephalitis or related disorders whose samples were sent for analysis at Centre de Référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, for anti-neural antibody study and then stored at the biobank Neurobiotec
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
HLA in autoimmune encephalitis and related disorders | 12 Months
  Description of HLA alleles and haplotypes carrier frequencies in autoimmune encephalitis and related disorders
Clinical relevance of HLA in autoimmune encephalitis and related disorders | 12 Months
  Description of clinical differences among patients regarding their HLA status

CONTACTS AND LOCATIONS:
Overall Officials: Jerome HONNORAT, PhD, Principal Investigator — Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes
Locations (1):
- Centre de référence des syndromes neurologiques paranéoplasiques et encéphalites auto-immunes, Lyon, France

IPD SHARING:
Plan to Share IPD: No